CLINICAL TRIAL: NCT06774300
Title: Evaluating Telehealth Delivery of Brief Alcohol Screening and Intervention for College Students
Acronym: Tele-BASICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of Houston (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Eric Pedersen, Associate Professor of Psychiatry and Behavioral Sciences, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA031252 (NIH); R01AA031252 (NIH)
Record Dates: First submitted 2024-12-31; First posted 2025-01-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Consumption
Keywords: alcohol; drinking; brief intervention; teleheath
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It will be clear to participants and facilitators which intervention condition participants are in. Therefore, masking will be conducted at the data analyses level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-person BASICS (Experimental): This intervention conditions consist of a feedback interview with a trained facilitator. The feedback interview is a one-hour intervention based on the information provided during the baseline assessment. The content and process of the interview will be similar to methods developed and tested by Marlatt and colleagues and described in detail in the BASICS manual. Trained facilitators will meet individually with the students in-person and provide concrete personalized feedback regarding the following BASICS content: drinking patterns, drinking norms, risks, beliefs about alcohol and its effects, and protective behavioral strategies
  Interventions: Behavioral: BASICS
- Tele-BASICS (Experimental): This intervention conditions consist of a feedback interview with a trained facilitator just like in the in-person BASICS condition. However, the feedback interview will be conducted over Zoom. Trained facilitators will meet individually with the students using video conferencing software and provide concrete personalized feedback regarding the following BASICS content: drinking patterns, drinking norms, risks, beliefs about alcohol and its effects, and protective behavioral strategies
  Interventions: Behavioral: BASICS
- Treatment as usual (Active Comparator): The control group for this study will receive the universities' online program that is typically given to students as a first line sanction. The program is informed by BASICS, but includes no facilitator, either in-person or online. It is primarily text-based with some graphics. It contains alcohol information (physiological reactions at specific blood alcohol levels, safe drinking tips, signs of alcohol poisoning), descriptions of alcohol laws and policies (on campus, minor in possession laws), campus and national resources (e.g., contact information for crisis hotlines and student counseling center), and personalized feedback (e.g., number of calories consumed via alcoholic drinks, money spent on alcohol).
  Interventions: Behavioral: Online alcohol programming

INTERVENTIONS:
Behavioral: BASICS — The intervention is the BASICS protocol outlined in the BASICS manual. It includes an online self-administered assessment and then delivery of a feedback session either in-person or over Zoom.
  Arms: In-person BASICS; Tele-BASICS
Behavioral: Online alcohol programming — This is a control intervention that is used as the first-line sanction for students at the two universities. It is an online program, informed by BASICS content, but contains no facilitator and is self-directed.
  Arms: Treatment as usual

SUMMARY:
This research study will test the efficacy of a telehealth version of the Brief Alcohol Screening and Intervention for College Students (BASICS), which is the gold standard prevention and intervention approach to target heavy alcohol use on college campuses across the United States.

DETAILED DESCRIPTION:
In this study, the researchers will evaluate the efficacy of a tele-BASICS approach utilizing the ZOOM application compared to in-person BASICS and a lower threshold treatment as usual intervention. Three hundred mandated and 300 volunteer students who report hazardous drinking will be recruited from two large universities and randomly assigned to a condition (in-person BASICS, Tele-BASICS, or treatment as usual). Follow-up assessments will occur 1-, 3-, 6-, and 12-months post-baseline. The significance of this research lies in the potential to maximize access to the highest standard of care by establishing support for easier access without sacrificing any central features of the traditional BASICS intervention. In addition, many universities pragmatically adapted existing in-person interventions to remote-telehealth approaches in response to the COVID pandemic but now have no scientific basis for determining whether transitioning back to in-person approaches would be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 26 years of age
* fluent in understanding English
* a registered student at one of the two intervention sites
* adequate internet capabilities to support video-conferencing
* access to a webcam, which is a standard features of most laptops, mobile devices, and desktops
* engage in binge drinking (i.e., 4 or more standard drinks in a sitting for women or 5 or more standard drinks in a sitting for men) at least once in the past month (for the volunteer sample only)
* experienced at least one negative alcohol-related consequence in the previous month (mandated students would meet this due to receiving an alcohol sanction)
* reports a score of 2 or higher on questions about a) interest in reducing their drinking, or b) interest in not increasing their drinking.

Exclusion Criteria:

* not meeting inclusion criteria or unwillingness to participate

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | Assessed over the course of 12 months
  Quantity and frequency of alcohol use in the past month (i.e., how many days drank and how many drinks per occasion). Assessed at baseline and then 1-, 3-, 6-, and 12-months post-baseline.
Alcohol-related consequences | Assessed over the course of 12 months
  Young Adult Alcohol Consequences Questionnaire assesses past month consequences from alcohol use. Higher scores indicate more endorsement of the 24 consequences (yes/no) items on the scale. Outcome assessed at baseline and then 1-, 3-, 6-, and 12-months post-baseline

SECONDARY OUTCOMES:
Completion rates | One time assessment at end of program, after 1 session is completed 1 to 2 weeks post-baseline
  We will evaluate completion rates of the each of the three programs tested in this study. This will be indicated by whether participants attended their scheduled BASICS session or fully completed their online treatment as ususal alcohol program

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Pedersen, Ph.D., Principal Investigator — University of Southern California; Clayton Neighbors, Ph.D., Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be uploaded to the NIAAA Data Archive (NIAAADA) consistent with NIAAA protocols and requirements. Data will be shared to the repository for other researchers to access in non-identifiable form. Participants will be informed that their anonymous data will be uploaded to the NIAAADA.